CLINICAL TRIAL: NCT00417729
Title: Phase 4 Study Evaluation of the Effects of Acarbose Versus Glibenclamide on Mean Amplitude of Glycemic Excursions and Oxidative Stress in Patients With Type 2 Diabetes Insufficiently Controlled by Metformin
Brief Title: Effects of Acarbose Versus Glibenclamide on MAGE and Oxidative Stress in Patients With Type 2 DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Changhua Christian Hospital (Other)
Responsible Party: Wayne H-H Sheu, M.D., Ph.D., Taichung Veterans General Hospital, Taichung, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB951004/C06211
Record Dates: First submitted 2007-01-01; First posted 2007-01-04 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Acarobse; Metformin; oxidative stress; Mean amplitude Glycemic Excursion; Meal test
MeSH Terms: conditions — Diabetes Mellitus | interventions — Acarbose; Glyburide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- acarbose, glibenclamide (Active Comparator): acarbose vs. glibenclamide (background metformin therapy)
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Acarbose — After an 8-week period of metformin monotherapy (500 mg t.i.d.), all patients were randomised to add on either acarbose or glibenclamide. The doses of acarbose and glibenclamide were 50 mg t.i.d. and 2.5 mg t.i.d., respectively, for 4 weeks and force-titrated to 100 mg t.i.d. and 5 mg t.i.d., respectively, for the last 12 weeks.
  Other Names: glibenclamide

SUMMARY:
To compare effect of acarbose versus glibenclamide treatment on mean amplitude of glyclemic excursion and oxidative stress in diabetes individuals who failed to control their glucose by metformin therapy alone

DETAILED DESCRIPTION:
This is a randomised and open-label study conducted in 2 medical centers in central part of Taiwan. Type 2 diabetic outpatients were eligible if they were aged 30-70 years, were on mono- or dual oral antidiabetic drugs for at least 3 months, and had a glycated hemoglobin (HbA1c) value between 7.0% and 11.0%. Patients who were treated with insulin or drugs that promote weight loss, had impaired renal (serum creatinine concentration greater than 132.6 μmol/l) or liver (AST or ALT 2.5 times upper limit of normal range) function, had a history of hemoglobinopathy or chronic anemia, or women of child-bearing potential without adequate contraception were excluded. All patients provided their informed consent before they were enrolled in this study.

After an 8-week period of metformin monotherapy (500 mg t.i.d.), all patients were randomised to add on either acarbose or glibenclamide. The doses of acarbose and glibenclamide were 50 mg t.i.d. and 2.5 mg t.i.d., respectively, for 4 weeks and force-titrated to 100 mg t.i.d. and 5 mg t.i.d., respectively, for the last 12 weeks. A complete 72 hours of glucose monitoring using a continuous glucose monitoring (CGM) system and meal tolerance test (MTT) after a 10-h overnight fasting were performed before randomisation and in the end of study. Morning urine samples were collected for measurement of 8-iso prostaglandin F2α (8-iso PGF2α), a commonly used parameter of oxidative stress (13-14). The primary objectives are the changes of MAGE obtained from CGM and urinary excretion rate of 8-iso PGF2α. The secondary objectives include changes of HbA1c, lipid profiles including total cholesterol, low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), and triglycerides, oxidized low-density lipoprotein (ox-LDL), high-sensitivity C-reactive protein (hs-CRP), total adiponectin, and high-molecular weight (HMW) adiponectin.

ELIGIBILITY:
Inclusion Criteria:

* Patients may be included in the clinical trial only if they meet all of the following criteria:

  1. Male or female outpatients;
  2. Age 30 - 70 years;
  3. Patients have failed to achieve glycemic control with diet, exercise and max. 2 OHA; Hemoglobin A1c level between 7.0 to 11.0 % at V1 and 7-11.5 % at V4.
  4. Diagnosis of diabetes mellitus is over a minimum 3-month period;
  5. All patients give written informed consent;
  6. For female patients of childbearing potential, the following criteria will be applied:
* Using adequate contraception since last menses and will continue to use adequate contraception during the clinical trial.
* Not lactating.
* Negative pregnancy test (urine) within 7 days prior to the first dose of study medication. (Note: the inclusion criterion 6 does not apply to menopausal female).

Exclusion Criteria:

* Patients will be excluded from the clinical trial for any of the following reasons:

  1. Patients with a serum creatinine concentration greater than 132.6 mmol/L (1.5 mg/dL) or liver function impairment (AST and ALT 2.5 times upper limit of normal range);
  2. Patients have laboratory test abnormality (biochemistry, hematology, or urinalysis), which in the investigator's opinion might confound the clinical trial. However, patients with hyperlipemia, elevated cholesterol or triglyceride levels, or lipid metabolism disorders are eligible;
  3. Use of chronic insulin therapy;
  4. Patients with medical conditions that could promote lactic acidosis, such as renal or hepatic disease, unstable angina, congestive heart failure (New York Heart Association Functional Classification III and IV), or chronic obstructive pulmonary disease, e.g. respiratory insufficiency, hypoxemic condition;
  5. Patients with a history of hypersensitivity to metformin hydrochloride, glibenclamide or acarbose;
  6. Patients receive an investigational drug within 30 days prior to admission to the clinical trial;
  7. Patients with significant alcohol, drug or medication abuse as judged by the investigator.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Mean Amplitude Glycemic Excursion | before randomisation and end of study
  A Medtronic MiniMed Continuous Glucose Monitoring System (Northridge, CA) was used for continuous glucose measurements on an ambulatory basis for 72 consecutive hours and MAGE calculated from the dataset.
Oxidative stress | before randomisation and end of study
  Spot urine was collected for measurement of 8-iso PGF2 alpha excretion rate.

SECONDARY OUTCOMES:
HbA1c | before randomisation and end of study
  Glycated hemoglobin for evaluation of efficacy of glycemic control.
fasting glucose | before randomisation and end of study
  after an overnight fasting
Insulin response | before randomisation and end of study
  Evaluation by meal tolerance test. Patients were asked to consume 1.5 cans of Ensure Liquid (266 kcal/can, caloric contribution: 64% carbohydrate, 14% fat, and 22% protein) after a 10-h overnight fasting. Blood samples were drawn at 0, 10, 20, 30, 60, 90, 120, and 180 minute relative to the meal ingestion for the measurements of glucose and insulin.
Fasting lipids | before randomisation and end of study
  after an overnight fasting
hsCRP | before randomisation and end of study
  high-sensitivity C-reactive protein
oxLDL | before randomisation and end of study
  oxidized low-density lipoprotein
Adiponectin | before randomisation and end of study
  Total and high-molecular weight adiponectin

CONTACTS AND LOCATIONS:
Overall Officials: Wayne H Sheu, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Chen PH, Tsai YT, Wang JS, Lin SD, Lee WJ, Su SL, Lee IT, Tu ST, Tseng YH, Sheu WH, Lin SY. Post-meal beta-cell function predicts the efficacy of glycemic control in patients with type 2 diabetes inadequately controlled by metformin monotherapy after addition of glibenclamide or acarbose. Diabetol Metab Syndr. 2014 May 31;6:68. doi: 10.1186/1758-5996-6-68. eCollection 2014. PMID 24932223
- [Derived] Wang JS, Lin SD, Lee WJ, Su SL, Lee IT, Tu ST, Tseng YH, Lin SY, Sheu WH. Effects of acarbose versus glibenclamide on glycemic excursion and oxidative stress in type 2 diabetic patients inadequately controlled by metformin: a 24-week, randomized, open-label, parallel-group comparison. Clin Ther. 2011 Dec;33(12):1932-42. doi: 10.1016/j.clinthera.2011.10.014. Epub 2011 Nov 10. PMID 22078152